CLINICAL TRIAL: NCT07110493
Title: Study of Visual Perception Phenomena: Phosphene Mapping Induced by TMS and Its Relationship With Eye Movements
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skolkovo Institute of Science and Technology (Other)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Skoltech-N15
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Visual Snow Syndrome; Color Blindness; Healthy Volunteer
MeSH Terms: conditions — visual snow syndrome; Color Vision Defects | interventions — Transcranial Magnetic Stimulation; Electroencephalography; Eye-Tracking Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Visual Snow Syndrome (Experimental): Participants diagnosed with Visual Snow Syndrome according to ICHD-3 criteria. This group will undergo TMS, EEG, and eye-tracking to study the mechanisms of visual perception.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Electroencephalography (EEG); Device: Eye-Tracking
- Color-blind Participants (Experimental): Participants with a confirmed diagnosis of color blindness. This group will undergo TMS, EEG, and eye-tracking to compare visual processing with other groups.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Electroencephalography (EEG); Device: Eye-Tracking
- Healthy controls (Active Comparator): Healthy volunteers with no history of neurological, psychiatric, or visual disorders. This group serves as a baseline to compare the findings from the experimental arms.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Electroencephalography (EEG); Device: Eye-Tracking

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Single-pulse TMS is applied to specific areas of the visual cortex to non-invasively induce the perception of phosphenes (brief flashes of light). Stimulation is delivered using a TMS device, with the operator controlling the intensity and frequency parameters to a level equal to the phosphene-evoking threshold. During stimulation, participants are seated comfortably and asked to report the location of perceived phosphenes on a monitor and a physical grid, helping to map the cortical visual field.
Device: Electroencephalography (EEG) — Continuous brain electrical activity is recorded using a 128-channel gel-based EEG system (Skoltech). The EEG cap is fitted to the participant's head to capture neural responses with high temporal resolution throughout the session. The collected data is used to analyze brain activity changes, including the P300 component and other event-related potentials, to identify neural correlates of phosphene perception and the effects of TMS.
Device: Eye-Tracking — Eye movements are continuously monitored using a Tobii Defusion 2 eye-tracker (Skoltech) operating at 60 Hz. This device provides high-accuracy measurements of gaze fixation and saccades. Participants are instructed to fixate their gaze on one of five predetermined points on a screen (center, top, bottom, left, right), with the fixation point being determined randomly for each trial. The eye-tracking data is analyzed to assess the influence of gaze position on phosphene localization and to study any stimulation-induced changes in eye movement patterns.

SUMMARY:
The purpose of this basic science study is to better understand human visual perception. Phosphenes are flashes of light that can be induced using Transcranial Magnetic Stimulation (TMS). The location of these phosphenes is known to change with eye movements, but the exact influence of these movements is not fully understood.

The main questions this study aims to answer are:

How does stimulating specific areas of the visual cortex relate to where a person perceives a phosphene? How do eye movements affect the accuracy of mapping these sensations? The study will enroll three groups of adults (aged 18-65): patients with Visual Snow Syndrome, color-blind participants, and healthy volunteers.

During the experiment, participants will receive single-pulse TMS to their visual cortex. Simultaneously, their eye movements will be monitored with an eye-tracker, and their brain activity will be recorded with EEG. Participants will be asked to report the location of the perceived light flashes. This will help create a map of the brain areas responsible for visual sensations and clarify how eye movements influence this process.

ELIGIBILITY:
Inclusion Criteria:

For the "Patients with Visual Snow Syndrome" Arm:

Confirmed diagnosis of Visual Snow Syndrome according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria.

Presence of persistent, dynamic, tiny dots ("visual snow") across the entire visual field.

Presence of at least one of the following additional visual symptoms:

Palinopsia (prolonged afterimages). Photophobia (hypersensitivity to light). Nyctalopia (impaired night vision). Blurred vision. Patients whose symptoms appeared after a SARS-CoV-2 viral illness may be included.

For the "Color-blind Participants" Arm:

Presence of a color perception disorder. Must have a formal diagnosis of color blindness confirmed by specific ophthalmologic tests (e.g., Ishihara, Rabkin, Justova, or Stilling polychromatic plates, or the Farnsworth-Munsell test).

For the "Healthy Controls" Arm:

Absence of any active or past neurological, psychiatric, or ophthalmological disorders.

Exclusion Criteria:

General Criteria (Applicable to all participants):

Use of psychotropic drugs. Any contraindications to Transcranial Magnetic Stimulation (TMS), such as a history of epilepsy, seizures, or metallic implants in the head.

Pregnancy.

Specific to the "Patients with Visual Snow Syndrome" Arm:

Presence of any organic abnormalities in the eyes or visual system identified during a standard ophthalmologic examination.

Presence of comorbid psychiatric disorders or other medical conditions (e.g., migraine with aura) that could explain the symptoms.

Specific to the "Color-blind Participants" Arm:

Any non-congenital cases of color blindness. Presence of concomitant visual impairments that could affect visual perception independently of color blindness, such as cataracts, glaucoma, or macular degeneration.

Presence of concomitant neurological or psychiatric diseases, such as schizophrenia, epilepsy, or mood disorders, that could affect the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Topographic Map of Phosphene Localization | During the single study visit (session duration is 4 hours).
  Creation of a map showing the correlation between specific stimulated areas of the visual cortex and the reported location of perceived phosphenes in the visual field. The map is generated based on participant reports during TMS stimulation.

SECONDARY OUTCOMES:
Correlation between Eye Movements and Phosphene Localization | During the single study visit (session duration is 1-4 hours).
  Analysis of eye-tracking data to quantify the influence of gaze fixation points and saccadic eye movements on the reported location of TMS-induced phosphenes.
Change in Brain Activity measured by EEG | During the single study visit (session duration is 1-4 hours).
  Analysis of EEG data, including tensor analysis and the P300 event-related potential, to identify changes in brain activity and correlations with phosphene perception and localization.
Change in Psychomotor Performance | Baseline (before TMS session) and after the TMS session (approximately at 4 hours).
  Assessment of visual-motor coordination and attention levels measured by a psychomotor test. The test requires participants to track a moving target on a screen. Performance is measured by the number of errors (deviations from the target).

CONTACTS AND LOCATIONS:
Locations (1):
- Skolkovo Institute of Science and Technology (Skoltech), Moscow, Russia